CLINICAL TRIAL: NCT05801692
Title: Arterial Blood Gases in Weaning of Mechanical VEntilation
Acronym: WAVE
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: Centre Hospitalier Universitaire de Besancon (Other)
Responsible Party: Sponsor
Other Study IDs: CHUB WAVE
Record Dates: First submitted 2023-02-10; First posted 2023-04-06 (Actual); Last update posted 2023-04-06 (Actual); Status verified 2023-01

CONDITIONS: Weaning of Mechanical Ventilation

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Procedure: Weaning of mechanical ventilation — Weaning of mechanical ventilation is the time when the patient is ready for separation from ventilatory support until breathing without invasive support

SUMMARY:
Weaning of mechanical ventilation is an important phase of ICU (Intensive Care Unit) patient hospitalization. Patients have to pass a spontaneous breathing trial, can have a phase of pause with mechanical ventilation before extubation and then can be weaned of invasive mechanical ventilation. Spontaneous breathing trial can be performed with a T-Tube or with Pressure support without PEEP (End Expiratory Positive Pressure) . Duration of spontaneous breathing trial range from 30 minutes to 120 minutes. Some clinicians performed an arterial blood gases at the end of the spontaneous breathing trial but this practice is not really defined and clearly explained in recommendations. Patients can benefit of ventilation support after extubation like non invasive pressure support or high flow nasal canulae. The procedure can be very different from a center to another, especially for arterial blood gases at the end of spontaneous breathing trial. Our aim is to observe in a multicenter study the daily practice of weaning of mechanical ventilation especially for arterial blood gases.

ELIGIBILITY:
Inclusion Criteria:

* Older than 18 years
* first attempt of weaning of mechanical ventilation

Exclusion Criteria:

* withholding of life sustaining therapies
* spontaneous breathing trial unsuccessful

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients hospitalized in intensive care unit with invasive mechanical ventilation, first attempt of weaning of mechnical ventilation
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2022-12-21 (Actual); Primary Completion 2023-07-01 (Estimated); Study Completion 2023-10-01 (Estimated)

PRIMARY OUTCOMES:
Type of spontaneous breathing trial performed | In the 24 hours of spontaneous breathing trial
  Spontaneous breathing trial is performed either with pressure support or with a T-Piece

SECONDARY OUTCOMES:
Arterial blood gases at the end of spontaneous breathing trial | In the hour of spontaneous breathing trial
  Arterial blood gases are sometime performed at the end of the spontaneous breathing trial during weaning of mechanical ventilation. Spontaneous breathing trial takes from 30 to 120 minutes
Duration of spontaneous breathing trial | The day of the spontaneous breathing trial
  Duration in minutes
Ventilatory procedure at the end of spontaneous breathing trial: either immediate extubation or pressure support ventilation with intubation | The day of extubation if extubation performed
  the procedure at the end of spontaneous: the patient is either extubated immediately or benefit of about one hour of invasive pressure support with the settings before spontaneous breathing trial until extubation. Procedure of extubation is differed of about one hour.
Frequency and type of ventilatory support after extubation | The day of extubation if extubation performed
  Ventilatory is either not performed or if performed, with pressure support or high flow oxygen nasal canulae
Need for reintubation | During the seven days following extubation
  Reintubation is the need to reintubate the patient because of extubation failure
Etiology of reintubation | During the seven days following extubation
  The cause of reintubation (pulmonary edema, infectious pulmonary disease...)
Death | The first 28 days following extubation
  If the patient died
Ventilator associated pneumoniae | From 48 hours after extubation until extubation
  Pneumoniae acquired after more than 48 hours of mechanical ventilation
days alive without mechanical ventilation | during the first 28 days of intensive care hospitalization.
  The number of days without invasive mechanical ventilation support during the first 28 days of intensive care hospitalization.

CONTACTS AND LOCATIONS:
Locations (1):
- BARROT, Besançon, France

IPD SHARING:
Plan to Share IPD: No